CLINICAL TRIAL: NCT06558136
Title: Evaluation of Salivary Interleukin-6, Interleukin-8 and LIGHT Protein Levels in Individuals With Different Periodontal Conditions
Brief Title: Evaluation of Salivary Biomarker Levels in Individuals With Different Periodontal Conditions
Status: Completed | Type: Observational
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Doruk Sagsoz, Research Assistant of Periodontology, Izmir Katip Celebi University
Other Study IDs: 2024--SAEK-0040
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Periodontitis; Gingivitis; Periodontal Health
Keywords: periodontitis; gingivitis; periodontal health; IL-6; IL-8; LIGHT; salivary level
MeSH Terms: conditions — Periodontitis; Gingivitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Unstimulated saliva samples collected for biomarker analysis (without DNA extraction) will be retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Periodontium: Full-mouth clinical periodontal measurements recorded and saliva obtained.
  Interventions: Diagnostic Test: Saliva obtaining
- Gingivitis: Full-mouth clinical periodontal measurements recorded and saliva obtained.
  Interventions: Diagnostic Test: Saliva obtaining
- Periodontitis: Full-mouth clinical periodontal measurements recorded and saliva obtained.
  Interventions: Diagnostic Test: Saliva obtaining

INTERVENTIONS:
Diagnostic Test: Saliva obtaining — The patient was asked to sit upright and tilt his/her head forward to collect saliva samples. İn this way, unstimulated saliva was allowed to accumulate in the floor of the mouth. The accumulated saliva was collected in a sterile container. It was then transferred to a propylene tube. The tubes were centrifuged and the clear part at the top of the tube was taken with a sterile syringe and transferred to a different propylene tube with 0.5 ml in each tube. Tubes were stored at -80ºC until the day of analysis.

SUMMARY:
In order to determine the pathogenesis of chronic inflammatory diseases, the levels of various cytokines are examined in tissues and fluids taken from the body. Recent publications have investigated the role of Interleukin-6 (IL-6), Interleukin-8 (IL-8) and LIGHT in chronic inflammatory diseases. The aim of this study was to evaluate the levels of these cytokines in the saliva of healthy individuals with gingivitis and periodontitis and to investigate whether they are reliable biomarkers for the diagnosis of periodontitis.

In the current study, all oral clinical parameters of 60 systemically healthy individuals (20 healthy, 20 with gingivitis and 20 with periodontitis) who were admitted to the clinic for routine periodontal control will be measured and saliva samples will be taken from the patients. IL-6, IL-8 and LIGHT (biomarkers emphasizing inflammation in saliva samples) will be determined by enzyme-linked immunoassay (ELISA). Then, statistical analyses will be performed to interpret the difference in cytokine levels between the groups and the relationship between these cytokines and clinical parameters.

Possible significant differences between cytokine levels will reveal that these proteins and enzymes can be utilized as a diagnostic tool in periodontal diseases, to distinguish periodontal disease status from healthy, or as a guide for treatments.

DETAILED DESCRIPTION:
The aim of this clinical study is to comparatively examine the levels of IL-6, IL-8 and LIGHT Protein in saliva samples obtained from periodontally healthy individuals with gingivitis and periodontitis who presented to the clinic for routine periodontal controls. In line with the results obtained; it is planned to determine the potential of these biochemical mediators to be used as a diagnostic marker in the diagnosis of periodontal disease.

Periodontitis is a multifactorial disease involving 10-15% of the world's adult population, developing due to microbial dental plaque and characterized by loss of clinical attachment and destruction of connective tissue and alveolar bone. If left untreated, it causes inflammation to penetrate into deeper tissues and alter bone homeostasis, leading to tooth loss.

Gingivitis is an inflammation of the gingiva that does not cause destruction in the surrounding tissues surrounding the tooth and is characterized by edema in the gums and bleeding in more than 10% of all areas in the mouth. According to the 2017 Classification of Periodontal Diseases, gingivitis is divided into two as dental plaque-related gingivitis and non-dental plaque-related gingivitis. Gingivitis is often painless and rarely spontaneous bleeding is observed and for these reasons, individuals may recognize the disease late. Therefore, early diagnosis of gingivitis is important to prevent the transformation of gingivitis into periodontitis characterized by progressive bone destruction and connective tissue destruction.

Studies have shown that there are more than 700 bacteria with the ability to colonize in the human oral cavity, but an average of 200 to 300 bacterial species in an individual's mouth. Among these bacteria, there are bacteria associated with gingival health, such as Porphyromonas gingivalis (Pg), Tannerella forsythensis (Tf), and Treponema denticola (Td), which are called red complex bacteria; Fusobacterium nucleatum (Fn) subspecies, Prevotella intermedia (Pi) and Aggregatibacter actinomycetemcomitans (Aa), which do not belong to any group, have been associated with active tissue destruction and periodontitis disease progression.

It has been shown that pathogenic bacteria affect the host immune response rather than direct inflammatory bone and connective tissue destruction. One of the important points in the pathogenesis of periodontal disease is cytokines, a member of the acquired immune system. Studies have shown that the amount of proinflammatory cytokines such as interleukin-6 (IL-6), IL-8, interleukin-1 (IL-1) tumor necrosis factor- α (TNF-α) increase in blood plasma, saliva and gingival groove fluid.

LIGHT protein (TNFSF-14), a member of the tumor necrosis factor superfamily (TNFSF), is mostly secreted by T cells and immature dendritic cells, but it is also secreted by cells with immunological roles such as monocytes, granulocytes, splenocytes and spleen cells. LIGHT can bind HVEM and three membrane-bound TNFSF signaling receptors, namely lymphotoxin beta receptor (LTβR) and DcR3. LIGHT-LTβR binding has been shown to induce apoptosis. While HVEM is expressed on endothelial, dendritic, natural killer, T and B cells, LTβR is expressed on fibroblasts, monocytes, endothelial, epithelial and stromal cells. The interaction of LIGHT protein with HVEM or LTβR results in Nuclear-Factor-kappaB activation and ultimately cytokine production. It has also been shown that LIGHT protein can costimulate the T cellular response via HVEM, including CD4+ and CD8+ T cells.

Rheumatoid arthritis is a chronic, destructive inflammatory disease. Proinflammatory cytokines such as IL-1, TNF-a, matrix metalloproteinase (MMP-8, MMP-9) are increased in rheumatoid arthritis as well as in periodontitis . For these reasons, there are similarities between the immunopathogenesis of periodontitis and rheumatoid arthritis. In a study conducted in rheumatoid arthritis patients, LIGHT protein was shown to be an important proinflammatory biomarker positively correlated with bone destruction and statistically increased bone destruction. In another study conducted in patients with rheumatoid arthritis, serum levels of LIGHT protein were evaluated and it was shown that increased levels of LIGHT increased RANKL-dependent osteoclastogenesis and increased osteoclast formation independently of RANKL. Another conclusion from this study is that LIGHT protein may play a role in immunopathogenic conditions associated with local and systemic bone loss.

In another study conducted in rheumatoid arthritis patients, LIGHT increased the inflammatory response in synovial fibroblast cells and was suggested to be a new anti-cytokine therapy target for the treatment of rheumatoid arthritis .

In a study conducted in patients with multiple myeloma bone disease, LIGHT was shown to increase osteoclastogenesis; inhibit osteoblastic proteins osteocalcin, bone sialoprotein and osterix formation; and inhibit sclerostin osteoblastogenesis from monocytes.

In a study by Fan et al. , it was investigated whether LIGHT protein is a potential inflammatory biomarker. In 566 patients, LIGHT protein was shown to increase 16-fold in blood serum in the presence of pneumonia, an inflammatory disease.

Type 2 diabetes mellitus is characterized by dysregulation of carbohydrate, lipid and protein metabolism and is caused by impaired insulin secretion from pancreatic islet cells, insulin resistance or a combination of both. Studies have shown periodontitis as the 6th complication of diabetes mellitus and a positive two-way correlation has been proven. In a study conducted in patients with type 2 diabetes mellitus, it was shown that LIGHT protein showed dysfunction in pancreatic islet cells, increased inflammatory cytokine secretion and increased inflammatory response formation in endothelial cells.

In a study conducted in patients with multiple myeloma bone disease, LIGHT was shown to increase osteoclastogenesis; inhibit the formation of osteoblastic proteins osteocalcin, bone sialoprotein and osterix; and inhibit sclerostin osteoblastogenesis from monocytes investigated whether LIGHT protein is a potential inflammatory biomarker. In 566 patients, it was shown that LIGHT protein increased 16-fold in blood serum in the presence of pneumonia, an inflammatory disease.

Type 2 diabetes mellitus is characterized by dysregulation of carbohydrate, lipid and protein metabolism and is caused by impaired insulin secretion from pancreatic islet cells, insulin resistance or a combination of both . Studies have shown that periodontitis is the 6th complication of diabetes mellitus and a positive two-way correlation has been proven. In a study conducted in patients with type 2 diabetes mellitus, LIGHT protein was shown to show dysfunction in pancreatic islet cells, increased secretion of inflammatory cytokines and increased inflammatory response in endothelial cells.

The starting point of this current study was a study published in 2024 that examined proinflammatory cytokines in the gingival groove fluid after periodontal surgery and aimed to find a potential new biomarker. According to this study, LIGHT was shown to stimulate the formation of proinflammatory cytokines IL-6 and IL-8 and MMP-9 in human gingival fibroblasts and to be associated with increased periodontal pocket probing depth formation at 12 months after surgery. It has been suggested that LIGHT protein causes tissue destruction in human gingival fibroblast cells, causes tissue loss in soft tissue and bone, and contributes to the development of periodontitis. In this study, it was emphasized that more studies are needed to evaluate the relationship between LIGHT and periodontitis.

Interleukin-6 is a multifunctional cytokine defined as a B-cell differentiation factor involved in the maturation of antibody-producing cells. IL-6 is a single-chain protein produced by T cells, B cells, monocytes, fibroblasts and some other cell types . IL-6 can transmit signals to cells in two ways: conventional receptor-dependent signaling and trans signaling associated with the soluble IL-6 receptor. One of the most important systemic effects of IL-6 is the induction of an acute phase response. This acute phase response is the induction of proinflammatory cytokine production and stimulation of neutrophil chemotaxis. It also increases C-reactive protein (CRP) levels, the most common acute phase protein in humans. It also has properties such as increasing T cell activation and differentiation and increasing macrophage differentiation.

IL-6 also increases endothelial cell proliferation, leading to IL-8 and monocyte chemoattractant protein secretion. As a result of these processes, it causes leukocytes to come to the site of inflammation. It also increases the secretion of proinflammatory MMP enzymes together with Interleukin-1.

In a study, the effect of non-surgical initial treatment on IL-6 levels in healthy and periodontitis patients was examined. According to the results of this study, baseline gingival groove fluid IL-6 levels were found to be significantly higher in periodontitis patients than in healthy patients. After non-surgical periodontal treatment, a statistically significant decrease in IL-6 levels was observed. This study suggests that IL-6 may be a biomarker that can be used in the diagnosis of periodontitis.

In a study conducted in rats, it was shown that inhibition of IL-6 secretion in the setting of experimental periodontitis halted the proinflammatory activity induced by IL-6 and reduced alveolar bone resorption and decreased RANKL production.

In a cross-sectional study, IL-6 and IL-8 levels in saliva and gingival groove fluid obtained from healthy individuals and individuals with periodontitis were analyzed. In the results, IL-6 and IL-8 levels were found to be higher in both saliva and gingival groove fluid in patients with periodontitis than in healthy patients.

IL-8 is a proinflammatory chemokine and its expression is primarily regulated by activator protein and nuclear factor-kappa β-mediated transcriptional activity . IL-8 expression has been shown to be regulated by stimuli such as TNF-α, IL-1β, steroid hormones, including inflammatory signals. IL-8 has been characterized on the basis of its chemotactic activity and its ability to cause degranulation of human neutrophils. In vitro, it has two main effects: chemotaxis and release of granule enzymes. It acts as a chemoattractant and neutrophil activator for cytokines at inflammatory sites and can be secreted by endothelial cells, gingival fibroblasts, monocytes, neutrophils and phagocytes. The secretion of IL-8 facilitates the migration of neutrophils from highly vascularized gingival tissue to the gingival groove . IL-8 is the earliest secreted proinflammatory cytokine from gingival epithelial cells stimulated by pathogenic bacteria such as P. Gingivalis and T. Forsythia and can persist for as long as one week after secretion.

In a literature review study, it was emphasized that the number of IL-8 levels increased significantly in the presence of periodontitis, but more studies are needed due to different results in various studies. In another literature review study, it was emphasized that IL-8 serum level may be a potential biomarker in the evaluation of periodontitis, but more studies are needed.

According to the above information, there is no study in the literature evaluating IL-6, IL-8 and LIGHT levels in saliva samples in terms of periodontal disease. This current study aimed to investigate the changes of these cytokines in the presence of periodontal disease by comparatively examining IL-6, IL-8 and LIGHT levels in saliva samples obtained from periodontally healthy individuals with gingivitis and periodontitis, to show their potential to be used in the diagnosis of disease or to provide preliminary information for future treatments that may be performed through these cytokine pathways.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy participants.
* At least twenty permanent teeth present in the oral cavity.
* Non-smokers.
* No medication for continuous use.
* Not pregnant or breastfeeding.

Exclusion Criteria:

* Any oral or systemic disease.
* Regular use of systemic medications.
* Pregnancy or lactation.
* Received periodontal treatment within the last 6 months.
* Use of antibiotics, anti-inflammatory medications, or systemic corticosteroids in the last 6 months.
* Smokers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult individuals aged 18 to 70 years, including periodontally healthy subjects, patients with gingivitis, and patients with periodontitis, recruited from patients presenting for routine dental examinations at the Department of Periodontology, İzmir Katip Çelebi University
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Salivary LIGHT level | 24 hours after taking the clinical measurements at the first visit
  Total amount of LIGHT protein in saliva
Salivary IL-6 level | 24 hours after taking the clinical measurements at the first visit
  total amount of interleukin-6 in saliva
Salivary IL-8 level | 24 hours after taking the clinical measurements at the first visit
  Total amount of interleukin-8 in saliva

SECONDARY OUTCOMES:
Periodontal Probing Depth | during the the initial visit
  With the help of a periodontal probe, the distance between the gingival margin and the sulcus/pocket base will be measured from six points of the tooth: mesiobuccal, midbuccal, distobuccal, mesiopalatinal/lingual, mid buccal/palatinal and distobuccal/palatinal. During the measurement, care will be taken to ensure that the probe is parallel to the long axis of the tooth and that excessive force is not applied. The values will be summed and divided by 6 to calculate the average SCD for each patient.
Clinical Attachment Level | during the the initial visit
  With the help of a periodontal probe, the distance between the enamel-cement border and the sulcus/pocket base will be measured at six points of the tooth: mesiobuccal, midbuccal, distobuccal, mesiopalatinal/lingual, mid buccal/palatinal and distobuccal/palatinal. The values will be summed and divided by 6 to calculate the average amount of clinical attachment level for each patient.
Plaque Index | during the the initial visit
  For Silness&Löe plaque index measurement, values will be obtained from four surfaces of each tooth: mesial, distal, vestibular and palatinal. The values will be summed and divided by four to determine the PI score for each tooth. Scoring will be done as follows; 0: No bacterial plaque on the gingival area of the tooth surface.
  1. No bacterial plaque is visible on the surface of the tooth by eye, but after probing, bacterial plaque is observed at the tip of the probe.
  2. The gingival area is covered with a thin to moderate amount of bacterial plaque, which is visible by eye.
  3. There is a large amount of soft debris, the thickness of which completely fills the gingival groove and the interdental space is filled with soft debris.
Gingival Index | during the the initial visit
  According to Löe&Silness gingival index; vestibule, lingual, mesial and distal surfaces of all teeth will be examined. The values will be summed and divided by four to determine the GI score for each tooth.
  0: Healthy gingiva.
  1. Mild inflammation, mild discoloration and edema but no bleeding after probing.
  2. Moderate inflammation, edema, redness and brightness, bleeding on probing.
  3. Severe inflammation and redness, edema, ulceration and tendency to spontaneous bleeding.
Bleeding on probing | during the the initial visit
  The following index criteria will be used to determine the degree of inflammation in the soft tissue surrounding the vestibular, lingual, mesial and distal surfaces of all teeth. The number of positive (+) scoring areas on the examined surfaces will be calculated as a percentage of the total number of examined areas.
  (-): No bleeding when the periodontal probe is passed along the gingival sulcus. (+): Bleeding is present at the gingival margin.

CONTACTS AND LOCATIONS:
Overall Officials: Şükrü Enhoş, Study Director — Izmir Katip Celebi University, Faculty of Dentistry, Department of Periodontology
Locations (1):
- Izmir Katip Çelebi University Department of Periodontology, Izmir, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No